CLINICAL TRIAL: NCT05732558
Title: Assessment of Operative Time, Precision, and Safety of an Augmented Reality Navigation System (Endosight) for the Guidance of Bone Biopsy
Brief Title: Augmented Reality Navigation System (Endosight) for the Guidance of Bone Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R.A.W. - S.R.L. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ESBB1
Record Dates: First submitted 2023-01-16; First posted 2023-02-17 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Bone Lesion; Bone Tumor; Bone Infection
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Intervention Model Description: The study is designed to compare a prospective arm composed of 8 patients who were prescribed a CT-Guided bone biopsy (with the aid of endosight navigation system) with a retrospective arm with a bone lesion for which a percutaneous biopsy has been performed from January 2011 to May 2022 (without endosight navigation system)
Who Masked: Outcomes Assessor
Masking Description: all sensitive data regarding enrolled patients will be transmitted to the Outcomes Assessor anonymously (code assigned to the patient)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prospective (Experimental): 8 Patients who were prescribed a CT-guided percutaneous bone biopsy, performed with the aid of endosight navigation system
  Interventions: Procedure: 8 Patients who were prescribed a CT-guided percutaneous bone biopsy, performed with the aid of endosight navigation system
- retrospective (No Intervention): 8 Patients with a bone lesion for which a percutaneous biopsy has been performed from January 2011 to May 2022

INTERVENTIONS:
Procedure: 8 Patients who were prescribed a CT-guided percutaneous bone biopsy, performed with the aid of endosight navigation system — The study is based on a comparison of the number of CT scans required for needle placement in bone biopsies (trunk area) performed with augmented reality navigation system (endosight) and without.
  Other Names: augmented reality; endosight; Bone biopsy; Bone tumor; Bone Lesion
  Arms: prospective

SUMMARY:
The goal of this clinical study is to evaluate the duration of the procedure, the precision (distance between the needle tip and the centre of the target), and the safety of endosight system in the guidance for bone biopsies.

DETAILED DESCRIPTION:
In this study results obtained in the prospective group will be compared with those obtained in the retrospective group.

Total N° of patients: 16

PROSPECTIVE GROUP (treated WITH the guidance of endosight):

N° of patients: 8

RETROSPECTIVE GROUP (treated WITHOUT the guidance of endosight):

N° of patients: 8

Main objective of the study:

Reduction of execution times by at least 10 minutes; Reduction of the number of CT scans by at least 2 scans.

N°of hospitals involved: 2.

Duration: maximum 6 months from the date of the first enrollment.

No follow-up is expected.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a bone lesion for which a percutaneous biopsy is indicated;
* Informed consent signed by the patient for participation in the study.

Exclusion Criteria:

* Age < 18 years;
* Pregnant and lactating women (assessed through auto declaration of the patient)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Procedure time | During bone biopsy procedure (after the bone sample has been collected)
  Change in the total duration of the procedure (calculated from the time of local anesthesia injection to the time of bone sample collection)
Total number of CT-SCAN | During bone biopsy procedure (after the bone sample has been collected)
  Change in overall number of CT scans performed during the procedure (calculated as the total number of CT scans required to reach the target; from the 1° CT-scan (local anesthesia) to the last CT-scan (sample collection from the bone)

SECONDARY OUTCOMES:
endosight accuracy | During bone biopsy procedure (after the bone sample has been collected)
  Distance between the tip of the needle and the center of the target (from 0mm to 10mm)
Total radiation dose | During bone biopsy procedure (after the bone sample has been collected)
  Change in the total radiant dose received by the patient (calculated by summing the radiation emitted for each CT-Scan performed from the anesthesia-point to the collection-point)
Operator satisfaction | During bone biopsy procedure (after the bone sample has been collected)
  satisfaction level of the operator (from 0 to 5 - 1: poor satisfaction, 5: high satisfaction)
Side effects | During bone biopsy procedure (after the bone sample has been collected)
  Total number of major+minor side effects, reported during the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Galeazzi - Sant'Ambrogio, Milan, MI, Italy

REFERENCES:
- [Derived] Albano D, Messina C, Gitto S, Chianca V, Sconfienza LM. Bone biopsies guided by augmented reality: a pilot study. Eur Radiol Exp. 2023 Jul 20;7(1):40. doi: 10.1186/s41747-023-00353-w. PMID 37468652